CLINICAL TRIAL: NCT04183062
Title: A Phase 2 Study of the Safety and Efficacy of BIO-11006 in the Treatment of Recurrent Osteosarcoma and Ewing's Sarcoma in Patients With Lung Metastases
Brief Title: BIO-11006 for Osteosarcoma and Ewing's Sarcoma Lung Metastases
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The drug for this study was not available by the manufacturer. No patients enrolled.
Sponsor: Nicklaus Children's Hospital f/k/a Miami Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019023
Record Dates: First submitted 2019-11-11; First posted 2019-12-03 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Osteosarcoma Metastatic; Ewing's Sarcoma Metastatic
Keywords: bone cancer; sarcoma; lung metastases; pediatric cancers
MeSH Terms: conditions — Bone Neoplasms; Sarcoma | interventions — Drug Therapy; Gemcitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Chemotherapy plus BIO-11006 (Experimental): Patients will receive BIO-11006 in addition to GemTax chemotherapy. The BIO-11006 inhalation solution will be given by mouth inhalation twice daily. BIO-11006 will be given during the first three cycles of GemTax and then will be stopped. Subjects will continue with GemTax treatment for three additional cycles. If the patient shows lung progression (either clinical or on imaging) at any point after cycle 4 has been given, but had shown at least a partial response during the tumor assessment after cycle 3, BIO-11006 may be re-started at the discretion of the investigator and continued for the duration of the GemTax treatment.
  Interventions: Drug: Chemotherapy (gemcitabine & docetaxel) plus BIO-11006

INTERVENTIONS:
Drug: Chemotherapy (gemcitabine & docetaxel) plus BIO-11006 — BIO-11006 will be administered at a dose of 75 mg twice daily for patients over 5 years of age and under 18 years of age or 125 mg twice daily for patients 18 years of age or older. The study drug will be administered twice daily by nebulizer over 20 minutes.
  GemTax will be administered in 21-day cycles. Gemcitabine will be administered at a dose of 900 mg/m2 IV over 90 minutes on days 1 and 8. Docetaxel will be administered at a dose of 75 mg/m2 IV over 60 minutes on day 8.

SUMMARY:
This is a Phase 2 study of an investigational drug, BIO-11006, for the treatment of lung metastases in pediatric patients with advanced osteosarcoma or Ewing's sarcoma. This study will enroll up to 10 patients aged between 5 and 21 at Nicklaus Children's Hospital in Miami, FL. Patients will receive BIO-11006 in addition to chemotherapy consisting of gemcitabine and docetaxel. This study will test the hypothesis that BIO-11006 will enhance the effect of the gemcitabine and docetaxel chemotherapy to treat lung metastases in osteosarcoma and Ewing's sarcoma.

DETAILED DESCRIPTION:
This is a Phase 2, controlled study of BIO-11006 peptide given in addition to Gemcitabine and Docetaxel (GemTax) in the treatment of patients with advanced osteosarcoma or Ewing's sarcoma with lung metastases. Patients will receive BIO-11006 in addition to GemTax chemotherapy, which is a current institutional treatment option for recurrent Osteosarcoma and Ewings's Sarcoma. The BIO-11006 inhalation solution will be given by mouth inhalation twice daily. BIO-11006 will be given during the first three cycles and then will be stopped. Patients will continue on GemTax for up to 6 additional cycles and will be clinically assessed before every cycle and have standard-of-care imaging assessments after cycle 3, 6 and 9. If the patient shows lung progression (either clinical or on imaging) at any point after cycle 4 has been given, but had shown at least a partial response during the tumor assessment after cycle 3, BIO-11006 may be re-started at the discretion of the investigator and continued for the duration of the GemTax treatment. Subjects will be followed for disease status during routine clinical follow-ups for 9 months post the end of study treatment. The trial will be conducted at a single site.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic verification of Ewing's sarcoma or osteosarcoma at original diagnosis or at relapse
2. Recurrence within one year of end of previous therapy
3. Presence of lung metastases
4. Osteosarcoma patients must be ineligible for curative surgery
5. Ability to take inhaled medication by nebulizer and be willing to adhere to the BIO-11006 regimen
6. Females of reproductive potential must have a negative pregnancy test at screening and must agree to use a method of highly effective contraception during study participation.
7. Males of reproductive potential must agree to the use of condoms or other methods to ensure effective contraception with partner
8. Stated willingness to comply with all study procedures and availability for the duration of the study
9. Provision of signed and dated informed consent form

Exclusion Criteria:

1. Previously treated and progressed on gemcitabine and docetaxel
2. Central Nervous System (CNS) metastases
3. Contraindication to gemcitabine or docetaxel
4. Known allergic reactions to components of BIO-11006
5. Use of medications that are primarily metabolized by cytochrome P450 isoenzymes
6. Treatment with another investigational drug within 8 weeks of enrollment.
7. Current pneumonia or idiopathic pulmonary fibrosis
8. Absolute Neutrophil Count (ANC) < 750 cells/mm3
9. Platelet count < 75,000 cells/mm3
10. Hemoglobin <8.0 g/dL
11. Creatinine clearance (CrCL) < 45 mL/min
12. Bilirubin > upper limit of normal (ULN) for age
13. AST and/or ALT >1.5 x ULN concomitant with alkaline phosphatase >2.5 x ULN
14. Organ transplant or bone marrow transplant recipient
15. Pregnancy or lactation
16. Current smoker or tobacco use within 3 months prior to enrollment
17. Any febrile illness or other severe illness within 2 weeks of enrollment
18. Known history of human immunodeficiency virus, hepatitis B, hepatitis C or tuberculosis

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2021-12-12 (Actual)

PRIMARY OUTCOMES:
Safety - Treatment-emergent adverse events (TEAEs) | Up to 16 months
  Frequency, type, severity, and duration of TEAEs. Sources of TEAEs may include spontaneous patient reports, results of physical examinations, and clinical laboratory measurements. Simple descriptive statistics of frequencies, centrality and variability will be utilized to tabulate and summarize TEAEs. If sufficient number of TEAEs will be captured, frequencies, duration and severity will be compared.

SECONDARY OUTCOMES:
Efficacy - Progression Free Survival (PFS) | Up to 16 months
  PFS will be measured from Cycle 1 Day 1 until occurrence of event (such as death, disease progression or end of study).

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo De Angulo, MD, Principal Investigator — Nicklaus Children's Hospital
Locations (1):
- Nicklaus Children's Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blackshear PJ. The MARCKS family of cellular protein kinase C substrates. J Biol Chem. 1993 Jan 25;268(3):1501-4. No abstract available. PMID 8420923
- [Background] Brown HK, Schiavone K, Gouin F, Heymann MF, Heymann D. Biology of Bone Sarcomas and New Therapeutic Developments. Calcif Tissue Int. 2018 Feb;102(2):174-195. doi: 10.1007/s00223-017-0372-2. Epub 2017 Dec 13. PMID 29238848
- [Background] Green TD, Park J, Yin Q, Fang S, Crews AL, Jones SL, Adler KB. Directed migration of mouse macrophages in vitro involves myristoylated alanine-rich C-kinase substrate (MARCKS) protein. J Leukoc Biol. 2012 Sep;92(3):633-9. doi: 10.1189/jlb.1211604. Epub 2012 May 23. PMID 22623357
- [Background] Grohar PJ, Janeway KA, Mase LD, Schiffman JD. Advances in the Treatment of Pediatric Bone Sarcomas. Am Soc Clin Oncol Educ Book. 2017;37:725-735. doi: 10.1200/EDBK_175378. PMID 28561686
- [Background] Hartwig JH, Thelen M, Rosen A, Janmey PA, Nairn AC, Aderem A. MARCKS is an actin filament crosslinking protein regulated by protein kinase C and calcium-calmodulin. Nature. 1992 Apr 16;356(6370):618-22. doi: 10.1038/356618a0. PMID 1560845
- [Background] Singer M, Martin LD, Vargaftig BB, Park J, Gruber AD, Li Y, Adler KB. A MARCKS-related peptide blocks mucus hypersecretion in a mouse model of asthma. Nat Med. 2004 Feb;10(2):193-6. doi: 10.1038/nm983. Epub 2004 Jan 11. PMID 14716307